CLINICAL TRIAL: NCT02793648
Title: Phase II, Double-blind, Randomized, 1-way Cross-over, to Investigate the Effectiveness of the Combination of Ascorbic Acid (Vitamin C) and Tocopherol (Vitamin E) Versus Placebo for the Treatment of Depressive Disorders in Elderly
Brief Title: Effectiveness of Ascorbic Acid and Tocopherol for Depression in Elderly.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yolanda de Diego Otero (Other)
Responsible Party: Sponsor-Investigator, Yolanda de Diego Otero, MSc. PhD, The Mediterranean Institute for the Advance of Biotechnology and Health Research
Organization: The Mediterranean Institute for the Advance of Biotechnology and Health Research (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PI-0290-2012
Record Dates: First submitted 2015-11-30; First posted 2016-06-08 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Depression
Keywords: Depression; Elderly
MeSH Terms: conditions — Depression | interventions — Ascorbic Acid; alpha-Tocopherol; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Ascorbic acid 200mg twice a day for twelve weeks Alpha tocopherol 200mg twice a day for twelve weeks
  Interventions: Drug: Ascorbic Acid; Drug: Alpha tocopherol
- Placebo (Placebo Comparator): colloidal Silica 200mg twice a day for twelve weeks
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: Ascorbic Acid — Two daily oral doses of 200mg of encapsulated vitamin C twice a day, administered at breakfast and dinner
  Other Names: Vitamin C
  Arms: Treatment
Drug: Alpha tocopherol — Two daily oral doses of 200mg of encapsulated vitamin E twice a day, administered at breakfast and dinner
  Other Names: Vitamin E
  Arms: Treatment
Drug: PLACEBO — Two daily oral doses of 200mg of encapsulated placebo, administered at breakfast and dinner
  Other Names: colloidal silica
  Arms: Placebo

SUMMARY:
The trial aims to treat depression. The incidence of major depression in the elderly accounts for between 3.6 and 4.8% and increases to 8 to 37.4% when depressive disorders in general is studied. Besides depression in the elderly presents with cognitive impairment, impaired physical and social functioning, and predisposes to suicide. These are patients who often have multiple conditions and be taking numerous psychopharmacological treatments which hinders further treatment. The clinical trial will analyze the improvement in neuropsychiatric symptoms through different instruments The Beck Depression Inventory (BDI), State-Trait Anxiety Inventory (STAI), Life Events (AV), World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0), Wechsler Memory Scale (WMS-III), Mini mental state examination (MMSE), Clinical Global Impression (CGI) and metabolic changes in the blood test measurements; after 12 weeks of antioxidant (Ascorbic acid and Tocopherol) treatment or placebo, and then after 24 weeks on active treatment with the antioxidant combination (Ascorbic acid and Tocopherol).

DETAILED DESCRIPTION:
Objective: To evaluate the effect of the combination of the antioxidant Ascorbic acid and tocopherol, as therapy of the depressive disorder in the elderly.

* Design: Pilot clinical trial, Phase II , 6-month randomized, double-blind placebo-controlled one-way crossover clinical trial, with two treatment periods of 12 weeks duration.
* Setting: Regional University Hospital, Malaga.
* Subjects: people older tan 55 years diagnosed with depression.
* Intervention: 50 participants randomly assigned, to receive antioxidant vitamins C (ascorbic acid) and vitamin E (d-alpha-tocopherol) once a day or placebo for 12 weeks double-blind. In Study Period 2, all participants receive (open) active treatment. Outcome measures: improvement in depressive symptoms. Plasma antioxidant status, also memory will be assessed by Wechsler Memory Scale (WMS-III), and cognitive improvement will be analyzed using Mini mental state examination (MMSE) at 0, 3, 6 months during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild or moderate depression by Mini International Neuropsychiatric Interview (MINI).
* Having more than 55 years old
* Have signed the informed consent document before starting the participation in the trial

Exclusion Criteria:

* Any advanced severe or unstable disease.
* Previous diagnose and / or presence of severe mental disorder.
* Risk of suicidal behavior.
* Any treatment regimen, including treatment with psychotropic drugs and / or anticonvulsant therapy that has not been stable for a period ≥ 4 weeks prior to randomization.
* Current treatment with more than two psychoactive medications, including medications for seizures control.
* Intake more than 100 mg of vitamin E or C a day in the last 4 months.
* Hypoprothrombinemia secondary to vitamin K deficiency
* Glucose 6-phosphate dehydrogenase deficiency (G-6-PD).
* Treatment with oral anticoagulants.
* Initiate or change the pharmacological or non-pharmacological interventions during the course of the trial.
* Allergy to the formula components (or excipient used)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms through Beck Depression Inventory (BDI) | 0,3, 6 months

SECONDARY OUTCOMES:
Change in anxiety through the State Anxiety Inventory (STAI-S) | 0, 3, 6 months
Change in the memory through the Wechsler Memory Scale (WMS-III) | 0, 3, 6 months
Change in cognitive impairment through MINI MENTAL STATE EXAMINATION (MMSE) | 0,3, 6 months
Change in the disease through the Clinical Global Impression (CGI) | 0,3, 6 months
Change in the individual level of functioning through the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | 0,3, 6 months
Change in the levels of blood oxidative stress through the antioxidant level | 0,3, 6 months

OTHER OUTCOMES:
Safety and tolerability analyzing the registered side effects | 0,3, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lucia M Perez-Costillas, MD PhD, Principal Investigator — Hospital Regional universitario de Malaga. UGC Salud Mental.
Locations (1):
- Psychiatric Service. Hospital Regional Universitario, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No